CLINICAL TRIAL: NCT04402983
Title: The Effectiveness of Telerehabilitation-Based Physiotherapy in COVID 19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Principal investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Telerehab_Covid19
Record Dates: First submitted 2020-05-22; First posted 2020-05-27 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-05

CONDITIONS: Covid19; Telerehabilitation; Physical Therapy
Keywords: exercise; videoconference
MeSH Terms: conditions — COVID-19; Motor Activity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Group (Experimental): Physiotherapy will be carried out by conducting online conference method. Program content; Respiratory exercise (chest breathing, diaphragmatic breathing, basal expansion exercises), Breath control training, Active breathing techniques cycle Light aerobic exercise Posture exercises Self walking
  Interventions: Other: Physiotherapy
- Control group (No Intervention): Information and exercise brochure will be provided

INTERVENTIONS:
Other: Physiotherapy — Program content Respiratory exercise (chest breathing, diaphragmatic breathing, basal expansion exercises), Breath control training, Active breathing techniques cycle Light aerobic exercise Posture exercises Self walking
  Arms: Telerehabilitation Group

SUMMARY:
Problems such as breathlessness, exercise intolerance and loss of peripheral muscle strength can be observed in individuals who have been diagnosed with COVID19 and have been discharged. In our study, it was aimed to investigate the effect of telerehabilitation physical therapy intervention to these cases by using videoconferencing method on the physical condition of the cases.

DETAILED DESCRIPTION:
Problems such as breathlessness, exercise intolerance and loss of peripheral muscle strength can be observed in individuals who have been diagnosed with COVID19 and have been discharged. In our study, it was aimed to investigate the effect of telerehabilitation physical therapy intervention to these cases by using videoconferencing method on the physical condition of the cases. The exercise program will be a total of 6 weeks, 3 days a week. Online access will be carried out synchronously by telephone or computer, and training sessions will not be recorded in order to protect patient personal information. The cases will be evaluated online at the beginning of the study and at the end of the 6-week exercise program. The selected evaluation parameters have been selected considering the ease of online application.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-75
* Being diagnosed with COVID19 and being discharged by being treated
* Having technological facilities suitable for telerehabilitation access

Exclusion Criteria:

* Any presence of comorbidity that may prevent them from exercising
* Not agreeing to be included in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Modified Medical Research Council Dyspnea Score | Baseline to 6 weeks
  The mMRC Dyspnea Scale is best used to establish baseline functional impairment due to dyspnea attributable to respiratory disease; tracking the mMRC over time or with therapeutic interventions is of less certain clinical utility.The severity of dyspnea is rated on a scale of 0 to 4. "O" means no dyspnea perception, "4" means severe dyspnea perception.
Timed up and go test | Baseline to 6 weeks
  The Timed "Up and Go" (TUG) Test measures, in seconds, the time taken by an individual to stand up from a standard arm chair (approximate seat height of 46 cm, arm height 65 cm), walk a distance of 3 meters (approximately 10 feet), turn, walk back to the chair, and sit down.
  Normal healthy elderly usually complete the task in 10 seconds or less. Very frail or weak elderly with poor mobility may take 2 minutes or more.
  Clinical guide: <10 seconds = normal <20 seconds = good mobility, can go out alone, mobile without a gait aid <30 seconds = problems, cannot go outside alone, requires a gait aid A score of more than or equal to 14 seconds has been shown to indicate high risk of falls.
Visual analog scale to assess the pain severity | Baseline to 6 weeks
  Visual analog scale to assess the pain on a horizontal, non-calibrated line of 100 mm, ranging from very low (0) to very high (100) score.
The Short Physical Performance Battery (SPPB) | Baseline to 6 weeks
  The Short Physical Performance Battery (SPPB) is comprised of 3 tasks: a standing balance test (side by side, semi-tandem and tandem), a 4-m habitual gait speed, and 5 sit to stand from a chair. Each task is scored (based on time) from 0-4 points. The total score is 12 points and this represents the highest performance. It can be easily performed at home via video conferencing
Visual analog scale to assess the fatigue severity | Baseline to 6 weeks
  Visual analog scale to assess the fatigue severity on a horizontal, non-calibrated line of 100 mm, ranging from very low (0) to very high (100) score.

SECONDARY OUTCOMES:
BECK depression inventory | Baseline to 6 weeks
  This is a 21-item self-assessment scale designed by Aaron Beck in 1961 to measure the risk and level of depression.
Saint George Respiratory Questionnaire | Baseline to 6 weeks
  The SGRQ ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Esra Pehlivan, PhD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences Turkey, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pehlivan E, Palali I, Atan SG, Turan D, Cinarka H, Cetinkaya E. The effectiveness of POST-DISCHARGE telerehabilitation practices in COVID-19 patients: Tele-COVID study-randomized controlled trial. Ann Thorac Med. 2022 Apr-Jun;17(2):110-117. doi: 10.4103/atm.atm_543_21. Epub 2022 Apr 19. PMID 35651892